CLINICAL TRIAL: NCT03458884
Title: Does a Cardiorespiratory Interval Training Program at Home Improve Post-stroke Fatigue?
Brief Title: Does Cardiorespiratory Interval Training Improve Post-stroke Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Anna Brandal, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-420-31M
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Fatigue
Keywords: Stroke; Fatigue; PROBE design; Cardiorespiratory fitness; Cardiorespiratory training
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Intervention Model Description: 1:1 prospective randomized open-label trial with blinded evaluators (PROBE-design)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiorespiratory interval training (Experimental): Cardiorespiratory interval training program on ergometer cycle, 30-40 minutes, 3 days a week for 8 weeks.
  Interventions: Other: Cardiorespiratory interval training
- Usual care (No Intervention): Usual ESD care including information about post-stroke fatigue, support and practical advice about how to identify and manage fatigue symptoms in daily tasks, such as the adaptation and prioritization of activities, physical activity and rest.

INTERVENTIONS:
Other: Cardiorespiratory interval training — A structured cardiorespiratory interval training program on an ergometer cycle 3 days a week for 8 weeks.
  Arms: Cardiorespiratory interval training

SUMMARY:
Post-stroke fatigue is common and negatively influences post-stroke recovery. Today, there is insufficient evidence how to treatment post-stroke fatigue. Our objective is to investigate if a structured cardiorespiratory interval training program added to the early supported discharge (ESD)-service results in relieved post-stroke fatigue and increased oxygen uptake.

This is a 1:1 prospective randomized open- label trial(Two-centre study) with blinded evaluators (PROBE-design) of 50 participants referred to ESD with study start at 4 (±1) weeks after discharge from the stroke unit. The intervention group (N=25) receives a structured cardiorespiratory interval training program on ergometer cycle, 30-40 minutes, 3 days a week for 8 weeks. The cardiorespiratory interval training program comprises of 4x4 minute interval, at 70 to 80% of peak heart rate, interrupted by 3 minutes active recovery.

The control group (N=25) receives usual ESD care. The primary outcome will be a shift in the Swedish Fatigue Assessment Scale before intervention (baseline) versus 8 weeks months after start of intervention in the intervention and control groups. Secondary outcomes include cardiorespiratory fitness, compliance, adherence and adverse events.

DETAILED DESCRIPTION:
Stroke is a major cause of disability among adults. After stroke, post-stroke fatigue is a common and negatively influences post-stroke recovery. Today, there is insufficient evidence how to treatment post-stroke fatigue. Post-stroke fatigue is considered to have a multifactorial cause and it is biologically plausible that fatigue might be related to physical deconditioning and reduced physical activity.

After stroke, functional limitations often lead to a reduction in physical activity, which in turn may lead to decline in cardiorespiratory fitness. Cardiorespiratory fitness is often measured as peak oxygen consumption, VO2peak. Studies have reported that physical activity and cardiorespiratory fitness is lower in stroke victims than gender- and aged-matched healthy individuals.

Intervention aimed to increased cardiorespiratory fitness has been highlighted as an important component in in stroke rehabilitation. Guidelines for physical activity and cardiorespiratory fitness following stroke recommend cardiorespiratory training 20-60 minutes, 3-7 days a week at 50-80% of maximal heart rate. Interval training (4 x 4 minutes) has showed to improve cardiovascular fitness at different patient groups, including Stroke.

Today, stroke unit and early supported discharge service (ESD) is recommended as an effective way to improve patient outcome and quality of care following stroke. The ESD service provides support and rehabilitation for the patients in their own environment and the rehabilitation is often focused on activities in daily living and mobility.

The objective of this study is to investigate if a structured cardiorespiratory interval training program added to the early supported discharge (ESD)-service results in relieved post-stroke fatigue and increased oxygen uptake. Furthermore, the study will explore whether it is feasible and safe for patients with post-stroke fatigue to perform a structured cardiorespiratory interval training program in their home environment.

Method/design

This is a 1:1 prospective randomized open-label trial (Two-centre study) with blinded evaluators (PROBE-design) comparing 8 weeks structured cardiorespiratory interval training program added to standard ESD care compared with standard ESD care alone in 50 patients with post-stroke fatigue.

Study participants

Consecutive stroke patients who receives stroke unit care followed by ESD-service at Umeå Stroke Center, University Hospital, Umeå, Sweden and Gävle hospital, Region Gävleborg, Sweden. A stroke physician will examine the patients 4 (± 1) weeks after discharge from the stroke unit. The patients fulfilling the eligibility criteria will receive oral and written information. Thereafter, the potential participants will be given at least 24 hours until they are asked for written informed consent.

After informed consent, an incremental cardiopulmonary exercise test will be performed on an ergometer cycle (pre-treatment test). The participants will also estimate post-stroke fatigue with the Swedish fatigue assessment scale (S-FAS).

Randomization

Participants (N=50) eligible for study participation according to inclusion and exclusion criteria will be randomly assigned to the intervention group(N=25) or the control group(N=25). The randomization procedure will be web-based using program Minim. Minimization will be used to create groups for intervention and control in order to stratify groups and ensure balance at study entry with respect to significant variables. The participants will be stratified according to sex, age and stroke severity (Modified Rankin Scale 0-1 vs ≥2).

Treatment

Stroke patients in the control group will receive usual ESD care including information about post-stroke fatigue, support and practical advice about how to identify and manage fatigue symptoms in daily tasks, such as the adaptation and prioritization of activities, physical activity and rest.

The participants in the intervention group will receive structured cardiorespiratory interval training program on an ergometer cycle. This is in addition to usual ESD care. The training will be conducted 30-40 minutes, 3 days a week for 8 weeks. Based on the incremental cardiopulmonary exercise test (pre-treatment test) an individual training heart rate range of 70 to 80% of maximal heart rate (HR peak) will be set. The participants will wear a heart rate monitor during the training and be instructed to exercise within the heart rate range. An experienced physiotherapist will be present and guide the training sessions during the first weeks. When the participants become more familiar with the exercise, the physiotherapist will monitor the training through phone or telemedicine equipment.

. The training session will start with a 10 minutes warm-up followed by 25 minutes of 4x4 minute interval, at 70 to 80% of peak heart rate, interrupted by 3 minutes active recovery and 5 minutes cool down. In order to get a estimation of perceived exertion, the participant will rate on The Borg Rating of Perceived Exertion (RPE) scale every minute during the 4-minute intervals.

Statistical analysis

The sample size was estimated by a power calculation. The power calculation was based on the level of fatigue assessed with the Swedish Fatigue Assessment scale (primary outcome). The absolute reliability for the Swedish Fatigue Assessment scale is 9 points, which means that a 9 points change is required to indicate a real change of fatigue level. 21 persons per group are needed for power of 80 % significance level of 0.05 (2 sided t-test, assuming a standard deviation of 10). This calculation is based on a t-test assuming a standard deviation of 10 points. A total of 50 participants (25 participants per group) will enter this study. The analyses of primary and secondary outcome will be on the basis of intension to treat. Two-sided students t-test or two-sided Wilcoxon signed rank test will be used to compare groups for the pre-treatment test and post treatment test.

ELIGIBILITY:
Inclusion Criteria:

* Preliminary or final diagnosis of acute stroke due to Brain infarction: large vessel disease, lacunar syndrome, cryptogenic stroke Intracerebral hemorrhage
* Post-stroke fatigue (defined as a summation score of 28 or more on the S-FAS)
* Medical stability
* Independent living in Umeå or Gävle (in the nearby surrounding areas) and able to cycle an ergometer cycle.

Exclusion Criteria:

* Patients with severe stroke with modified Rankin Scale >3
* Atrial fibrillation, pacemaker or other arrhythmia which exclude reliable monitoring of heart-frequency
* Unstable pulmonary or cardiac disease
* Serious co-morbidity with for example terminal cancer, hemodialysis, severe cognitive dysfunction with Montreal Cognitive Assessment (MOCA) ≤ 26
* Drug abuse
* Patients living far away from the hospital or in residential care facilities.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Post-stroke fatigue | The S-FAS will be measured before intervention (pre-treatment test) and immediately after end of 8 week intervention (post-treatment test)
  Post-stroke fatigue will be measured with The Swedish Fatigue Assessment Scale (S-FAS) comprises 10 questions that describe how a person generally feels. The answers are given using a 5-point scale ranging from 1 (never) to 5 (always) such that the total score ranges from 10 to 50 points. Items 4 and 10 require reversed scoring. A high score indicate an increase level of fatigue.

SECONDARY OUTCOMES:
Cardiorespiratory fitness (Peak oxygen consumption, VO2peak) | Cardiorespiratory fitness (peak oxygen consumption) will be measured before intervention (pre-treatment test) and immediately after end of 8 week intervention (post-treatment test)
  Cardiorespiratory fitness will be determined by measuring peak oxygen consumption (VO2peak) in an incremental cardiopulmonary exercise test on a ergometer cycle
Feasibility (Fidelity) | Fidelity will be measured throughout the intervention and will be monitored at each individual training session, 3 days a week for 8 weeks
  Fidelity will be measured by recording the number of sessions completed.
Feasibility (Adherence) | Adherence will be measured throughout the intervention and will be monitored at each individual training session, 3 days a week for 8 weeks
  Adherence will be measured by monitoring heart rate (HR) during the exercise
Feasibility (Adverse events) | Adverse events will be measured throughout the intervention and will be monitored at each individual training session, 3 days a week for 8 weeks
  Adverse events will be recorded by asking the participants to fill in a home-exercise logbook at each training session and reviewing hospital record.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bråndal, PhD, Principal Investigator — Department of Community Medicine and Rehabilitation, Physotherapy
Locations (1):
- Anna Bråndal, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No